# Statistical Analysis Plan Addendum

**Study Title:** A phase I/II study of lutetium (177Lu)-lilotomab satetraxetan

(Betalutin®) antibody-radionuclide-conjugate for treatment

of relapsed non-Hodgkin lymphoma.

**Version:** Final 1.0 (30 May 2022)

Nordic Nanovector Study No: LYMRIT-37-01 PART A – Phase I & IIa

Syne qua non Study No: NOR18001

### For Syne qua non Ltd – Lead Statistician

DocuSigned by:

Elaine Howarth

Signer Name: Elaine Howarth

Signing Reason: I am the author of this document Signing Time: 30-May-2022 | 4:08:45 PM BST

-1165E56AC9F04FF2885587ACA0901BE0

### For Nordic Nanovector

DocuSigned by:

Christine Wilkinson Blanc

U

Signer Name: Christine Wilkinson Blanc Signing Reason: I approve this document Signing Time: 30-May-2022 | 2:30:53 PM PDT

-331B8876519845F8B86862BB2763BF42

Date:30MAY2022 Version: Final 1.0

# **Table of Contents**

| L | List of Abbreviations | 3 |
|---|-----------------------------------------------------|----|
| N | Modification History | 4 |
| | 1 Introduction | |
| 2 | 2 Dose Limiting Toxicity | 5 |
| | 2.1 Existing Text | 5 |
| | 2.2 Reason and Justification for Addendum | 5 |
| | 2.3 Strategy for analysing DLTs | 7 |
| 3 | 3 Haematological Episode | 9 |
| | 3.1 Existing Text | 9 |
| | 3.2 Reason and Justification for Addendum | 9 |
| | 3.3 Strategy for analysing Haematological Episodes | 9 |
| 4 | 4 Disease History | 10 |
| | 4.1 Existing Text | 10 |
| | 4.2 Reason and Justification for Addendum | 10 |
| | 4.3 Inclusion of additional Disease History Outputs | 11 |


### List of Abbreviations

CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events

DLT Dose Limiting Toxicity
FL Follicular Lymphoma

MedDRA Medical Dictionary for Regulatory Authorities

PT Preferred Term

SAP Statistical Analysis Plan SOC System Organ Class

SRC Safety Review Committee

TEAE Treatment Emergent Adverse Event

TFL Tables, Figures and Listings

Date:30MAY2022

# **Modification History**

| Version | Change History | Reason | Date |
|---------|----------------|--------|-----------|
| 1.0 | First Version | N/A | 30MAY2002 |

Date:30MAY2022 

### 1 Introduction

This addendum to the Statistical Analysis Plan (SAP) version 5.0 (dated 05APR2022) describes necessary clarifications to the Dose Limiting Toxicity (DLT) and Haematological Episodes analyses to be conducted for the LYMRIT-37-01 Phase I/IIa study (Part A). It also includes a small addition to the disease history analyses for Phase IIa Follicular Lymphoma (FL) patients.

This addendum must be read and applied in conjunction with the finalised and approved SAP version 5.0 (dated 05APR2022) for LYMRIT-37-01 Phase I/IIa (Part A) and the Table, Figure and Listing (TFL) Shells version 6.0 (dated 06APR2022).

## **2** Dose Limiting Toxicity

### 2.1 Existing Text

In section 3.13.2 of the SAP version 5.0 (dated 05APR2022), a DLT is defined as follows:

A Dose Limiting Toxicity (DLT) will be confirmed for a Phase I participant following a clinical review by the sponsor of the following data:

### Haematological:

- 1. A haematological parameter with a grade 4 toxicity recorded post-baseline that does not recover to grade 3 within 7 days.
- 2. A TEAE term of PT = "THROMBOCYTOPENIA" or "FEBRILE NEUTROPENIA" or "PLATELET COUNT DECREASED" or any PT containing either "HAEMORRHAGE" or "BLEEDING".

### Non-haematological:

• A serum biochemistry parameter with a grade 3 toxicity or more.

Confirmed DLT AEs from study Day 1 to Day 92 (Month 3) will be summarised by SOC and PT for Phase I only).

All confirmed DLTs for Phase I participants only will be summarised.

All confirmed DLTs will be listed (for Phase I only) detailing date recorded, whether haematological or non-haematological, the laboratory parameter (where applicable), the laboratory value (where applicable), the toxicity grade (where applicable) and the adverse event detail (where applicable).

### 2.2 Reason and Justification for Addendum

The criteria definitions for DLT used within the SAP version 5.0 (dated 05APR2022) are in line with LYMRIT-37-01 protocol version 11.0 (dated 27OCT2017) onwards.

The Phase I/IIa (Part A) participants on the LYMRIT-37-01 study provided informed consent to earlier versions of the protocol. As the protocol versions have evolved over the years, the DLT criteria definitions have also been revised and amended.

A summary of the change in DLT definitions between the various versions of the protocol is summarised below:

Date:30MAY2022 

# <u>LYMRIT-37-01 Protocol versions 4.0 to 7.0 inclusive</u> (4.0, 14Sep2012; 5.0, 25Mar2013; 6.0, 11Mar2014; 6.0B, 18Feb2015; 7.0, 26Nov2015)

Dose Limiting Toxicity was defined as:

Dose limited toxicity (DLT): Toxicity will be graded according to CTCAE version 4.

- Haematologic DLT is defined as grade 4 haematological toxicity that does not recover after 7 days, or grade 3 haematological toxicity that does not recover after 2 weeks.
- Non-haematologic DLT defined as grade 3 or more. However, the non-haematologic events will be evaluated by the safety review committee in the study and the decision will be taken by them to define whether the non-hematologic events are DLT or not.

### LYMRIT-37-01 Protocol version 8.0, 04Jul2016

Dose limiting toxicity for Phase 1 arm 1 was defined as the following:

Toxicity will be graded according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE; version 4).

- Haematologic DLT is haematology parameters defined as grade 4 that does not recover after 7 days, or grade 3 that does not recover after 2 weeks.
- Non-haematologic DLT defined as grade 3 or more, however, the non-haematologic events will be evaluated by the safety review committee in the study and decision will be taken by them to define whether the non-haematologic events are DLTs or not.

The safety review committee will make the recommendation whether to move to next dose level.

Dose limiting toxicity has been revised and is defined as the following for arms 2, 3, 4, 5 and phase II:

Haematology:

- Haematological grade 4 toxicity that does not recover to grade 3 within 7 days,
- or bleeding due to thrombocytopenia, or febrile neutropenia,
- or failure of platelets or neutrophils to recover to grade 1 by 12 weeks after treatment.

Non-haematological: grade 3 or more, final decision as to whether the non-haematological toxicity is a DLT will be made by the Safety Review Committee for this study.

### LYMRIT-37-01 Protocol version 9.0, 28Nov2016 & version 10.0, 04Jul2017

Dose limiting toxicity was defined as the following:

Haematology:

- Haematological grade 4 toxicity that does not recover to grade 3 within 7 days,
- or bleeding due to thrombocytopenia, or febrile neutropenia,
- or failure of platelets or neutrophils to recover to grade 1 by 12 weeks after treatment.

Non-haematological: grade 3 or more, final decision as to whether the non-haematological toxicity is a DLT will be made by the Safety Review Committee for this study.

Plus clarification of the following: The DLT criteria that previously applied to Arms 2, 3, 4, 5 and phase II will also apply to Arm 1 phase I patients, to harmonise the assessment of the safety data of all enrolled patients/treatment arms.

NB all patients enrolled in LYMRIT-37-01 Part A (Phases I and IIa), were enrolled under Protocol versions 4.0 to 10.0 inclusive.

Date:30MAY2022 

### LYMRIT-37-01 Protocol version 11.0, 27Oct2017

Dose Limiting Toxicity was defined as:

- Haematological:
- Grade 4 toxicity that does not recover to grade 3 within 7 days
- or bleeding due to thrombocytopenia, or febrile neutropenia
- Non-haematological:
- Grade 3 or more, final decision to be made by the SRC.

The DLT criteria were re-visited by the SRC in May 2017, and a recommendation was made to re-define "failure of platelets or neutrophils to recover to grade 1 by 12 weeks post-Betalutin" as not being a DLT event, as this is not associated with adverse clinical outcomes, is not a widely recognised hematologic DLT parameter in chemotherapy or RIT studies and is not aligned with the DLT criteria from other Betalutin studies.

### 2.3 Strategy for analysing DLTs

To account for the changes in the DLT definitions over the course of the study period for Phase I/IIa (Part A), the DLT definitions as outlined in Protocol Version 9.0 will be used for all participants irrespective of the Protocol version the participant was initially consented.

The Table below provides a summary of DLT criteria and related programming (NB this applies to time period from Day 1 to Week 12) for Phase I participants only:

| <b>Protocol Versions</b> | DLT Criteria | Programming Requirements |
|---|---|---|
| 4.0-7.0 Phase I Arm 1 Not applied due to re- evaluation under Version 9.0 | <ul> <li>Grade 4 haematological toxicity* that does not recover after 7 days</li> <li>Grade 3 haematological toxicity* that does not recover after 2 weeks.</li> </ul> | <ul> <li>Grade 4 haematology lab value that lasts ≥7 days</li> <li>Grade 3 haematology lab value that lasts ≥2 weeks</li> </ul> |
| | • ≥Grade 3 non-<br>haematological toxicity*<br>with review/decision by<br>SRC | <ul> <li>◆ ≥Grade 3 biochemistry lab value</li> <li>◆ Any Grade ≥3 AE PT except the following:</li> <li>◆ AE PT THROMBOCYTOPENIA</li> <li>◆ AE PT PLATELET COUNT DECREASED</li> <li>◆ AEPT NEUTROPENIA</li> <li>◆ AE PT NEUTROPHIL COUNT DECRESAED</li> <li>◆ AE PT ANAEMIA</li> <li>◆ AE PT LYMPHOPENIA</li> <li>◆ AE PT LYMPHOCYTE COUNT DECREASED</li> </ul> |
| 8.0-10.0<br>Phase I Arms 2, 3, 4, 5<br>and Phase IIa<br>Note: The Phase 1 Arm | Grade 4 haematological<br>toxicity* that does not<br>recover to grade 3 within 7<br>days | Grade 4 haematology lab value that lasts ≥7 days |
| 1 patients were re-<br>evaluated under Version<br>9.0 to these criteria | Bleeding due to<br>thrombocytopenia | <ul><li>Any one of the following AE PTs:</li><li>HAEMATURIA</li><li>EPISTAXIS</li></ul> |

Date:30MAY2022 

| | | <ul> <li>HAEMORRHAGE</li> <li>PT containing BLEEDING</li> <li>AND any one of the following concomitantly:</li> <li>AE PT THROMBOCYTOPENIA</li> <li>AE PT PLATELET COUNT DECREASED</li> <li>Grade 1 to 4 platelet laboratory value</li> </ul> |
|---|---|---|
| | Febrile neutropenia | AE PT FEBRILE NEUTROPENIA |
| | Failure of platelets or neutrophils to recover to grade 1 by 12 weeks after treatment. | • Any ≥Grade 2 value during the first 12 weeks that is not Grade 0 or 1 at Week 12 |
| | | <ul> <li>≥Grade 3 biochemistry lab value</li> <li>Any Grade ≥3 AE PT</li> </ul> |
| 11.0 onwards (not applicable for Part A as all patients were enrolled under versions 4.0 to 10.0 inclusive. Applicable to Part B/C only. | <ul> <li>Grade 4 haematological toxicity* that does not recover to grade 3 within 7 days</li> <li>Bleeding due to thrombocytopenia</li> <li>Febrile neutropenia</li> <li>≥Grade 3 non-haematological toxicity* with review/decision by SRC</li> </ul> | • As above |

<sup>\*</sup>Haematological toxicity = haemoglobin, neutrophils, lymphocytes and platelets only

The definition of 'confirmed DLT' in the SAP version 5.0 (dated 05APR2022) is superseded by the definition of programmatically derived DLT in the SAP addendum. A Dose Limiting Toxicity (DLT) will be confirmed for a Phase I participant following a clinical review by the sponsor of the programmatically derived data.

Programmatically derived DLT AEs from study Day 1 to Day 92 (Month 3) will be listed by SOC and PT for Phase I participants only.

All programmatically derived DLTs will be listed (for Phase I only) detailing date recorded, whether haematological or non-haematological, the laboratory parameter (where applicable), the laboratory value (where applicable), the toxicity grade (where applicable) and the adverse event detail (where applicable).

In cases, where the Safety Review Committee reviewed DLTs according to a version of the DLT definitions different from that present in the protocol version in place at the time the participant was initially consented, resulting discrepancies (if any) will be individually discussed in the Clinical Study Report for LYMRIT-37-01 Phase I/IIa (Part A).

In a change to the existing text in SAP version 5.0 (dated 05APR2022), all DLT AEs from study Day 1 to Day 92 (Month 3) will not be summarised by SOC and PT for Phase I only. This summary table is now to be omitted (reference: Table 14.3.2.1.1.A in the TFL shells version 5.0, dated 06APR2022) from the final outputs. As originally stated, all

Date:30MAY2022 

programmatically derived DLTs will be listed for Phase I only (reference: Listing 16.2.7.3.1.A in the TFL shells version 5.0, dated 06APR2022) in the final outputs.

## 3 Haematological Episode

### 3.1 Existing Text

In section 3.13.3 of the SAP version 5.0 (dated 05APR2022), a haematological episode is defined as follows:

For Phase IIa participants a haematological episode will be confirmed from the following data:

- 1. A haematological parameter with a grade 4 toxicity recorded post-baseline that does not recover to grade 3 within 7 days.
- 2. A TEAE term of PT = "THROMBOCYTOPENIA" or FEBRILE NEUTROPENIA" or "PLATELET COUNT DECREASED" or any PT containing either "HAEMORRHAGE" or "BLEEDING".

All confirmed haematological episodes for Phase IIa participants will be summarised and listed.

#### 3.2 Reason and Justification for Addendum

Regarding haematological episodes for the Phase IIa participants, the same reasoning and justification for the addendum regarding DLTs for Phase I participants is also applicable i.e. in that from Protocol Version 9.0, they harmonised the assessment of the safety data of all enrolled patients/treatment arms.

Therefore, the definition for haematology/haematological DLTs in Protocol version 9.0 will be applied when defining the criteria for haematological episodes experienced by Phase IIa participants.

### 3.3 Strategy for analysing Haematological Episodes

As with the DLTs, to account for the changes in the DLT definitions over the course of the study period for Phase I/IIa (Part A), the DLT definitions as outlined in Protocol Version 9.0 will be used for all participants irrespective of the Protocol version the participant was initially consented.

Haematological Episodes will be programmatically derived using haematology laboratory parameters and the definitions for DLT. The Table below provides a summary of Haematological episodes criteria and related programming (NB this applies to time period from Day 1 to Week 12) for Phase IIa patients only:

| <b>Protocol Versions</b> | Haematological episodes | Programming Requirements |
|---|---|---|
| 8.0-10.0<br>Phase I Arms 2, 3, 4, 5<br>and Phase IIa | • Grade 4 haematological toxicity* that does not recover to grade 3 within 7 days | Grade 4 haematology lab value that lasts ≥7 days |
| Note: The Phase 1 Arm 1 patients were re-evaluated under Version 9.0 to these criteria | Bleeding due to<br>thrombocytopenia | Any one of the following AE PTs: HAEMATURIA EPISTAXIS HAEMORRHAGE PT containing BLEEDING |

Date:30MAY2022 

| | • AND any one of the following |
|---------------|----------------------------------|
| | concomitantly: |
| | AE PT THROMBOCYTOPENIA |
| | AE PT PLATELET COUNT |
| | DECREASED |
| | Grade 1 to 4 platelet laboratory |
| | value |
| Febrile neutr | ropenia • AE PT FEBRILE |
| | NEUTROPENIA |

<sup>\*</sup>Haematological toxicity = haemoglobin, neutrophils, lymphocytes and platelets, only

The definition of 'confirmed' in the SAP version 5.0 (dated 05APR2022) is superseded by the definition of confirmed in the SAP addendum. A Haematological Episode will be confirmed for a Phase IIa participant following a clinical review by the sponsor of the programmatically derived data.

Programmatically derived Haematological Episode AEs from study Day 1 to Day 92 (Month 3) will be listed by SOC and PT for Phase IIa participants only.

In cases, where the Safety Review Committee reviewed haematological events according to a version of the haematological event definitions different from that present in the protocol version in place at the time the participant initially consented, resulting discrepancies (if any) will be individually discussed in the Clinical Study Report for LYMRIT-37-01 Phase I/IIa (Part A).

In a change to the existing text in SAP version 5.0 (dated 05APR2022), all programmatically derived Haematological Episodes from study Day 1 to Day 92 (Month 3) will not be summarised by SOC and PT. This summary table is to be omitted from the final outputs (reference: Table 14.3.2.1.2.A in the TFL shells version 5.0, dated 06APR2022). As originally stated, all programmatically derived haematological episodes will be listed for Phase IIa (reference: Listing 16.2.7.3.1.A in the TFL shells version 5.0, dated 06APR2022) in the final outputs.

# 4 Disease History

### **4.1 Existing Text**

In section 3.7.3 of the SAP version 5.0 (dated 05APR2022), it states the following:

"Disease history (initial diagnosis of NHL and current status of NHL) will also be summarised for the subgroup of FL participants only".

### 4.2 Reason and Justification for Addendum

For the disease history of the subgroup of Phase IIa FL participants, in addition to the initial diagnosis of NHL and current status of NHL being summarised for the subgroup of Phase IIa FL participants only, the Sponsor has also requested that the previous treatment for NHL and prior systemic therapies for NHL are also summarised for the subgroup of Phase IIa FL participants only.

Date: 30MAY2022 

### 4.3 Inclusion of additional Disease History Outputs

In a change to the existing TFL shells version 5.0 (dated 06APR2022) for the final outputs, two additional (repeated) tables will be included as follows:

- Table 14.1.5.1.A.4 Disease History Previous Treatment for Non-Hodgkin Lymphoma (NHL) Information Part A Phase IIa Patients with Follicular Lymphoma
- Table 14.1.5.2.A.4 Disease History Prior Systemic Therapies for Non-Hodgkin Lymphoma (NHL) Part A Phase IIa Patients with Follicular Lymphoma

Date:30MAY2022 

# **DocuSign**

### **Certificate Of Completion**

Envelope Id: 87990E7ECADA4136B5ADB4FE1CD9FF05

Subject: Please DocuSign: Statistical Analysis Plan Addendum - Final 1.0.docx

Source Envelope:

Document Pages: 11 Signatures: 2 Envelope Original Certificate Pages: 5 Initials: 0 Elaine Howarth

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Envelope Originator: Elaine Howarth 134 Turnpike Road Southborough, MA 01772

Elaine.Howarth@veristat.com IP Address: 20.68.172.95

Status: Completed

#### **Record Tracking**

Status: Original Holder: Elaine Howarth Location: DocuSign

| 30 May 2022 16:03 | Elaine.Howarth@veristat.com | , and the second |
|---|---|---|
| Signer Events | Signature | Timestamp |
| Christine Wilkinson Blanc<br>cwilkinsonblanc@phi-medics.co.uk<br>Security Level: Email, Account Authentication<br>(Required) | Signature Adoption: Pre-selected Style Signed by link sent to cwilkinsonblanc@phi-medics.co.uk Signature ID: 331B8876-5198-45F8-B868-62BB2763BF42 Using IP Address: 109.145.88.11 | Sent: 30 May 2022 16:08<br>Resent: 30 May 2022 16:11<br>Viewed: 30 May 2022 22:30<br>Signed: 30 May 2022 22:30 |
| | With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document | I |

#### **Electronic Record and Signature Disclosure:**

Accepted: 30 May 2022 | 22:30

ID: d3ce3611-1414-4680-9416-78e588d556ff

Elaine Howarth
elaine.howarth@veristat.com
Senior Statistician
Security Level: Email, Account Authentication

Elaine Howarth

Sent: 30 May 2022 | 16:08 Viewed: 30 May 2022 | 16:08 Signed: 30 May 2022 | 16:08

Signature Adoption: Pre-selected Style

Signed by link sent to elaine.howarth@veristat.com

Signature ID:

1165E56A-C9F0-4FF2-8855-87ACA0901BE0

Using IP Address: 20.68.172.95

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I am the author of this document

### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

(Required)

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |

| Certified Delivery Events | Status | Timestamp |
|---|---|---|
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Summary Events Envelope Sent | Status Hashed/Encrypted | <b>Timestamps</b> 30 May 2022 16:08 |
| • | | • |
| Envelope Sent | Hashed/Encrypted | 30 May 2022 16:08 |
| Envelope Sent<br>Certified Delivered | Hashed/Encrypted<br>Security Checked | 30 May 2022 16:08<br>30 May 2022 16:08 |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted Security Checked Security Checked | 30 May 2022 16:08<br>30 May 2022 16:08<br>30 May 2022 16:08 |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Veristat (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

### **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Veristat:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: vincent.hughes@veristat.com

### To advise Veristat of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at vincent.hughes@veristat.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from Veristat

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to vincent.hughes@veristat.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Veristat

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to vincent.hughes@veristat.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Veristat as described above, you consent to receive exclusively
  through electronic means all notices, disclosures, authorizations, acknowledgements, and
  other documents that are required to be provided or made available to you by Veristat
  during the course of your relationship with Veristat.